CLINICAL TRIAL: NCT04836754
Title: The Effect of Covid-19 on Breast Milk Microbiome and Its Bioactive Components
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Aysu Yıldız Karaahmet (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Sponsor-Investigator, Aysu Yıldız Karaahmet, PhD, Halic University
Organization: Halic University (Other)
Other Study IDs: Covid-19
Record Dates: First submitted 2021-04-07; First posted 2021-04-08 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Covid19; Human Milk
Keywords: covid-19; human milk; microbiota; microbiome; bioactive ingredient
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: Pregnant women with Covid-19
- Control groups: Pregnant women who do not have Covid-19

SUMMARY:
Coronavirus disease (Covid-19) is a new public health crisis threatening humanity caused by SARS-CoV-2. Although it originated in China's Hubei province in late 2019, it has spread to many countries around the world. Although Covid-19 first caused infection by affecting the lung, current data showed that the gastrointestinal tract was also affected by detecting viral RNA in Covid-19-infected human intestinal epithelial cells and feces. The association has been confirmed by showing that patients hospitalized with COVID-19 have significant changes in intestinal bacterioma. These changes have been characterized by a significant reduction in gut microbiome (BM) diversity associated with gastrointestinal complaints of the acute phase of infection (e.g. abdominal pain, nausea, vomiting, diarrhea), depletion of beneficial bacterial symbionts, and enrichment of opportunistic pathogens (e.g. Streptococcus, Rothia, Actinomyces). In particular, recent studies have evidence that patients with Covid-19 are more prone to a dysbiosis profile of the gut microbiota, infected individuals present irregular gut microbiota, and even dysbiosis (disruption of microbiota balance) in the gut microbiota.

The first case reports reported in China suggested that there was no virus found in amniotic fluid, umbilical cord blood, throat swabs of the newborn, placenta, vaginal fluid, and breast milk samples infected with Covid-19. The latest data indicate that there is no vertical transmission to the fetus, and so far, no viruses have been found in the cord blood of newborns born from Covid-19 positive pregnant women, nasal sampling and amniotic fluid and placentas of pregnant women. However, the effect of intestinal microbial structure affected by Covid-19 on breast milk microbiota and the effect of a dysbiosis to occur on infant health or the effect of the healing properties of breast milk on Covid-19 are still not clearly known. This views are that intestinal microbial colonization originating from the gastrointestinal system affected by Covid-19 will affect breast milk microbial colonization. However, there is no study on this subject.

For this purpose, aim in this study was to determine the breast milk microbiome and biologically active proteins (secretory immunoglobulin A (sIgA), lysozyme, lactoferrin, osteoprotegerin (OPG), leptin, adiponectin and β-endorphin (b-) levels of mothers who had Covid-19 with healthy mothers. will be compared.

DETAILED DESCRIPTION:
Coronavirus disease (Covid-19) is a new public health crisis threatening humanity caused by SARS-CoV-2. Although it originated in China's Hubei province in late 2019, it has spread to many countries around the world (Wang et al., 2020). In patients with Covid-19, severe cases of respiratory, hepatic, gastrointestinal and neurological complications and a complex clinical picture that eventually turns into death are observed (Guo et al., 2020; Li et al., 2020). The underlying pathophysiological mechanisms are complex and multifactorial, and have been summarized as a hyper-response of the immune system that causes an inflammatory / cytokine storm (Li et al., 2020).

Although Covid-19 caused infection by first affecting the lung, current data showed that the gastrointestinal system was also affected by detecting viral RNA in human intestinal epithelial cells and feces infected with Covid-19 (Cheng et al., 2002; Wu et al., 2020). This is thought to be caused by the relationship between the gut microbiota and the lung axis. Studies have demonstrated that Bacteroidetes and Firmicutes bacteria, which are dominant in intestinal colonization, are also dominant in the lung (Bacteroidetes, Firmicutes and Proteobacteria) (Zhang et al., 2020). In short, while intestinal microbiota causes lung diseases, respiratory tract virus infections also cause confusion in the intestinal microbiota. In fact, many studies have shown that respiratory infections are associated with a change in the composition of the gut microbiota (Groves et al., 2020). The high-throughput 16S rRNA amplicon sequence and shotgun metagenomic sequence analyzes demonstrated that hospitalized COVID-19 patients had significant changes in the intestinal bacterioma, and the relationship was confirmed. These changes have been characterized by a significant reduction in gut microbiome (BM) diversity associated with gastrointestinal complaints of the acute phase of infection (e.g. abdominal pain, nausea, vomiting, diarrhea), depletion of beneficial bacterial symbionts, and enrichment of opportunistic pathogens (e.g. Streptococcus, Rothia, Actinomyces) (Gu et al., 2020; Zuo et al., 2020). In particular, recent studies have evidence that patients with Covid-19 are more prone to dysbiosis profile of the gut microbiota, infected individuals present irregular gut microbiota and even dysbiosis (disruption of microbiota balance) in the gut microbiota (Gu et al., 2020; Zuo et al., 2020 ).

The intestinal flora plays a protective role in many metabolic and immune functions of the host, i.e. against pathogenic colonization of the virus, including training and strengthening the immune system to fight infections (Fernandes et al., 2019). Looking at the composition of the gut flora, it is highly dynamic from birth and is shaped by different environmental factors (e.g. diet, breast milk pre- / probiotics, drugs) resulting in various microbial-host functions (Koppel, Maini Rekdal, Balskus, 2017; Weiss, Hennet, 2017) . Human gastrointestinal tract (GIS), 2000 'classified into 12 different phyla, the most common (> 90%) Proteobacteria (Gram-negative), Firmicutes (Gram-positive), Actinobacteria (Gram-positive) and Bacteroidetes (Gram-negative) phyla. It is believed that human intestinal viroma, consisting of both prokaryotic and eukaryotic viruses, shares important information with all microbial components and can affect overall human health by shaping the structure and function of the intestinal community (Cani , 2018; Garmaeva et al., 2019).

Breast milk is the bioactive component that most affects the formation of neonatal microbial colonization in the postnatal period and provides us with information about human future health. Breast milk is not only the best nutritional source for babies, but it is also known to contain immune components such as secretory antibodies, immune cells, antimicrobial proteins (such as lactoferrin and lysozyme), cytokines, and human milk oligosaccharide. Before the 2000s, breast milk was thought to be sterile, and the presence of bacteria indicated contamination or infection. However, several researchers have shown that breast milk has been colonized with bacteria since pregnancy and contains commensal bacteria in particular. In a study, it was found that Proteobacteria (Gram-negative), Firmicutes (Gram-positive), Actinobacteria (Gram-positive) and Bacteroidetes (Gram-negative) phyla, which are dominant in maternal intestinal colonization, are among the breast milk microbes Firmicutes, Proteobacteria Bacteroidetes and Actinobacteria. It has been proved that breast milk originates from the mother's gastrointestinal system in this case (Ojo et al., 2018). In addition, the same study showed that there were bacteria sharing the same strains in the mother's intestine, the baby's intestine and breast milk, and the mother's commensal bacteria had vertical transmission to the infant's intestine through breast milk.

Human coronaviruses were defined as enveloped, positive-sensitive, single-stranded RNA viruses, first described in 1965 (Tyrrell and Bynoe, 1965). There are seven identified strains known to infect humans. Four of the strains (alphacoronaviruses 229E, NL63, OC43, and betacoronavirus HKU1) are ubiquitous in humans and cause the common cold. There are questions about the effect of human coronaviruses on pregnant, maternal and infant health and the transmission status is not clear. Pregnancy alters a woman's immune system and makes them more susceptible to infections. However, there is currently no evidence that pregnant women are more likely to be affected by COVID 19 or serious illness as a result, compared to the general population. Although the mechanism is unclear, there is limited evidence that one of the four strains (229E) mentioned above can be transmitted vertically from mothers to infants (Gagneur et al., 2008). The presence of this virus (229E) in neonatal gastric samples suggests that a possible mechanism for infection is through breast milk, but this study did not specifically evaluate breast milk (Gagneur et al., 2008).

The first case reports reported in China suggested that there was no virus in amniotic fluid, umbilical cord blood, throat swabs of the newborn, placenta, vaginal fluid, and breast milk samples infected with Covid-19 (Johns et al, 2013). The latest data indicate that there is no vertical transmission to the fetus, and so far, no viruses have been found in the cord blood of newborns born from Covid-19 positive pregnant women, nasal sampling and amniotic fluid and placentas of pregnant women. However, the effect of intestinal microbial structure affected by Covid-19 on breast milk microbiota and the effect of a dysbiosis to occur on infant health or the effect of the healing properties of breast milk on Covid-19 are still not clearly known. This study views are that intestinal microbial colonization originating from the gastrointestinal system affected by Covid-19 will affect breast milk microbial colonization. However, there is no study on this subject.

Breast milk is a golden nutrient that provides critical nutrients and bioactive compounds that support growth and immune development during infancy. Variation in milk components and bioactive compounds as a result of demographic and genetic factors, the mother's lifestyle and exposure has both positive and negative effects on infant health (Abrahamsson et al., 2009; de Andres et al., 2018; Johns et al. , 2013). It has been reported that babies who are breastfed have a dynamic gut microbiome and the incidence of some diseases has decreased (Abrahamsson et al., 2009; de Andres et al., 2018). In addition to macro and micronutrients and bioactive compounds, breast milk contains many types of bacteria. Lactoferrin is one of the important bioactive components in breast milk. The lactoferrin in breast milk can support a local intestinal environment, such as microbiota that strengthens the innate defenses of newborns. Lactoferrin promotes the growth of favorable gut microbiota and the proliferation of enterocytes through direct anti-inflammatory and immunomodulatory effects.

The action of lactoferrin on cell receptors prevents viral damage, surface accumulation and cell entry. In this way, it protects and strengthens mucosal immunity and intestinal epithelial barrier. It is believed that breast milk, particularly lactoferrin, exhibits potential antiviral effects. The challenge is how effective they are in preventing viral infections such as coronaviruses (de Andres et al., 2018).

We believe early breastfeeding provides vital prevention during viral outbreaks due to the high value of colostrum and breast milk and the specific role of lactoferrin, but more clinical evidence is needed. These effects and mechanisms have not been tested on Covid-19, but we can consider this approach as they affect other coronaviruses.

In addition, breast milk components containing approximately 109 bacteria are known to affect the baby's own microbiome and immune system (Ruiz et al., 2019). However, contrary to what is known, breast milk microbiota and its influencing factors are only recently being discovered and understood (McGuire & McGuire, 2017; Moossavi et al., 2019; Williams et al., 2017). In addition, while exploring the effects of certain components in breast milk on the nursing baby, we tend to ignore the dynamic state and effect of other components that could greatly affect the results. While it was known that the microbiome, which we cannot see with the naked eye, could affect individuals, it was not thought that our world would change that much with a single virus, Covid-19. While the microbiome we often ignore because it is invisible to us reminds us of a world that has profound effects on our health and well-being, how does Covid-19 affect this world and breast milk? For this purpose, aim in this study was to determine the breast milk microbiome and biologically active proteins (secretory immunoglobulin A (sIgA), lysozyme, lactoferrin, osteoprotegerin (OPG), leptin, adiponectin and β-endorphin (b-) levels of mothers who had Covid-19 with healthy mothers. will be compared.

A total of 20 mothers (10 mothers) and healthy (10 mothers) who had Covid-19 in the last month of pregnancy between April 2021 and June 2021 will be included in the study and the mothers will be given an appointment on the 15th day and will start with taking breast milk samples and 16sRNA microbiota. Analyzing the microbiota content of breast milk and the levels of biologically active proteins (secretory immunoglobulin A (sIgA), lysozyme, lactoferrin, osteoprotegerin (OPG), leptin, adiponectin and β-endorphin (b)) in breast milk content will be evaluated.

Hypothesis in this study is that breast milk microbiota will differ in variety and composition in mothers who have had Covid-19. In this direction, as a result of the research; Conducting microbial analysis to evaluate the content of microbiota and bioactive components by taking the milk of mothers who have had Covid-19 during pregnancy,

- In line with the results obtained, it is planned to give correct advice and guidance in accordance with an urgent problem.

ELIGIBILITY:
Inclusion Criteria:

* The cognitive level of the mother is sufficient to understand and answer the questions,

  * Having a single pregnancy,
  * Mother's ability to read, write and understand Turkish
  * The time of delivery is in the range of 37 <GH <42 weeks
  * Not having a chronic disease of the mother (Diabetes, hypertension, hypothyroidism etc.) Vaginal delivery
  * The mother's not using antibiotic derivative drugs during pregnancy
  * Getting 10 points below the Beck Depression Scale
  * Absence of prematurity, Introuterine Growth Retardation (IUGR) or genetic disease in the newborn
  * Birth weight in the range of 2500-4000 gr
  * Absence of a gastrointestinal disease in the newborn
  * Feeding more than 50% of the baby with breast milk
  * Absence of Premature Membrane Rupture (PROM) for more than 24 hours at birth

Exclusion Criteria:

* Expressing breast milk or having problems with the breast,
* The mother's use of probiotics before randomization and during pregnancy,
* The inclusion of sampled mothers in other clinical studies at the same time.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — mothers on the first day after birth
Study Population: The sample of the study: The population of the study will be 20 mothers who are hospitalized in the obstetrics clinic of the SBU Istanbul Sultangazi Haseki Training and Research Hospital for emergency delivery, who had Covid-19 during pregnancy (10 mothers) and healthy (10 mothers). Power analysis to determine the size, G-Power 3.1.9.2. program (Zuo et al., 2020). According to this calculation, a total of 20 mothers, a minimum of 10 mothers in each group, will be included in the sample, with a 95% confidence interval, alpha 0.05 and 80% power, with a 20% improvement difference between the two groups.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
data analysis:maternal and infant health | postpartum 15th day
  Data Collection Form, Quality of Life Scale
Microbiological Analysis:human milk | postpartum 15th day
  16sRNA analysis

CONTACTS AND LOCATIONS:
Overall Officials: Aysu Yıldız Karaahmet, Phd.Student, Principal Investigator — Halic University; Gülümser Dolgun, Profesor, Study Director — Istanbul University - Cerrahpasa; Ceren Ozkul Kocak, Asist prof, Study Director — Hacettepe University
Locations (1):
- Haseki Training and Research Hospital, Sultangazi, Istanbul, Turkey (Türkiye)